CLINICAL TRIAL: NCT03916549
Title: The Role of Traditional Acupuncture in Low Anterior Resection Syndrome Treatment - Pilot Study
Brief Title: Acupuncture in Low Anterior Resection Syndrome Treatment
Acronym: AcuLARS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other)
Collaborators: Vilnius University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AcuLARS
Record Dates: First submitted 2019-04-13; First posted 2019-04-16 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Low Anterior Resection Syndrome
MeSH Terms: conditions — Low Anterior Resection Syndrome | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: One group of intervention - acupuncture for LARS patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group 1 (Experimental): The patients with bowel dysfunction following low anterior resection performed at least 1 year ago will undergo acupuncture. The acupuncture procedure is performed by one well trained person, 1 time per week in total of 10 weeks on the same day time. Sterile, disposable, stainless steel acupuncture needles (40x0.25 mm diameter) were inserted to corporal acupoints, with initial gentle stimulation by quick rotation of 1080°, after then leaving needle in located place for twenty minutes. Needling deep - 0.5-1 cm. If the intent was to invigorate - the needle was inserted to the flow of energy; if harmonization needed - the needle was placed perpendicular to the point flow of energy; if sedation was needed, needles were placed against to the flow of energy on channel. The selection of acupoints was based according by traditional Chinese medicine, literature findings.
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — The acupuncture procedure is performed by one well trained person, 1 time per week in total of 10 weeks on the same day time. Sterile, disposable, stainless steel acupuncture needles (40x0.25 mm diameter) were inserted to corporal acupoints, with initial gentle stimulation by quick rotation of 1080°, after then leaving needle in located place for twenty minutes. Needling deep - 0.5-1 cm. If the intent was to invigorate - the needle was inserted to the flow of energy; if harmonization needed - the needle was placed perpendicular to the point flow of energy; if sedation was needed, needles were placed against to the flow of energy on channel. The selection of acupoints was based according by traditional Chinese medicine, literature findings.

SUMMARY:
Acupuncture has it's role in treating patients with fecal incontinence and diarrhea-predominant irritable bowel syndrome. There is no trial or case-report assessing it's role in treatment of Low anterior resection syndrome.

DETAILED DESCRIPTION:
Colorectal cancer is common in Western countries. For thirty years rectal cancer treatment is standardized: patients are undergoing low anterior resection with mesorectal excision +/- (chemo)radiotherapy. Unfortunately around 80% of patients undergoing low anterior resection will experience complex bowel dysfunction including fecal incontinence, soiling, urgency, incomplete evacuation, fragmented defecation and impaired rectal sensation known as low anterior resection syndrome (LARS) causing a "toilet dependence" which severely affects quality of life.

Still there is no standardized treatment for LARS.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 year
* signed written consent
* patients experiencing major low anterior resection syndrome
* patients at least one year following the surgery

Exclusion Criteria:

* allergy to stainless steal
* implanted pacemaker
* current skin infection
* needle phobia
* metastatic disease to the central nervous system (brain, spinal cord)
* at the same time, application of smecta, dicetel, cisapride or traditional Chinese medicine;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Bowel function changes after the treatment using Low anterior resection syndrome questionnaire | 6 months
  Bowel function assessment using Low anterior resection syndrome questionnaire Bowel function following low anterior resection surgery for rectal cancer will be assessed using Low anterior resection syndrome score (LARS score - simple 5 question questionnaire). LARS score is a tool consisting of five items, which are as follows: incontinence due to flatus (score range from 0 to 7), incontinence due to liquid stools (score range from 0 to 3), frequency of bowel movements (score range from 0 to 5), clustering (score range from 0 to 11) and urgency (score range from 0 to 16). The severity of each item is calculated on a scale ranging from 0 to 42, with a score of 0-20 (no LARS), 21-29 (minor LARS) and 30-42 (major LARS).

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Vilnius, Lithuania

REFERENCES:
- [Result] Dulskas A, Aukstikalnis T, Kavaliauskas P, Samalavicius NE. The Role of Traditional Acupuncture in Low Anterior Resection Syndrome Treatment: A Pilot Study. Dis Colon Rectum. 2022 Jan 1;65(1):93-99. doi: 10.1097/DCR.0000000000002060. PMID 34882631